CLINICAL TRIAL: NCT05917652
Title: THE Actuate-CBC Study: Accelerating the Uptake of Telemedicine for Crisis Burn Care
Brief Title: The Actuate-CBC Study
Acronym: ACTUATE
Status: Recruiting | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Amanda Bettencourt, Assistant Professor, University of Pennsylvania
Other Study IDs: 850877
Record Dates: First submitted 2023-01-20; First posted 2023-06-26 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Telemedicine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- RedCap surverys: The study team will use REDCap to send an IRB approved secure electronic survey
  Interventions: Behavioral: Tool kit
- Interviews: The study team plans to do about 18-23 one-on-one interviews with clinicians (burn care nurses, physicians, advanced practice providers, therapists) or will progress until data saturation is reached.
  Interventions: Behavioral: Tool kit

INTERVENTIONS:
Behavioral: Tool kit — The study team will develop and design key elements of the implementation intervention (toolkit) among a small group of burn and non-burn clinician stakeholders (4-6 total). The study team will use in-person interviews with stakeholders and a semi-structured interview guide to elicit feedback and assess face and content validity of the toolkit elements prior to deployment across the study hospitals. For those who consent to participation, the study team will conduct virtual teleconference interviews in-person using a secure videoconferencing platform while the person is not working, at a time convenient for them. Interviews will last between 45 and 60 minutes. The study team anticipates conducting 4-6 interviews to finalize toolkit elements prior to implementation.

SUMMARY:
The study team will use implementation science to accelerate the uptake of teleconsultationfor burn patients by 1) examining the relationships between clinician perceptions of acceptability, feasibility, intention to use, and actual use of burn teleconsultation 2) identifying the optimal process for burn teleconsultation and the barriers and facilitators for its use during a crisis or prolonged care situation, and 3) designing and testing the effectiveness of a specific, tailored burn teleconsultation toolkit intervention to increase burn teleconsultation use.

DETAILED DESCRIPTION:
The principal investigator's central hypothesis is that a tailored implementation intervention (toolkit) that integrates the known advantages of using telemedicine for burn consultation with new knowledge regarding clinician perceptions and the setting in which they work will improve the feasibility, acceptance, intention to use, and uptake of burn teleconsultation. The implementation intervention will enable rapid burn teleconsultation implementation under crisis circumstances and assist clinicians to virtually connect the person caring for a burn patient anywhere to the entire burn team's expertise. The study results will lead to more robust national crisis, wartime, and disaster response plans, improve quality of burn care, and decrease morbidity and mortality from serious burn injury, regardless of injury location.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older and
* are providing burn care to patients at the 4 burn centers and the non-burnhospitals are eligible for inclusion.

Exclusion Criteria:

* do not meet inclusion criteria,
* decline to participate or do not give consent to participate in the study, •
* directly express uneasiness about the participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: physicians and other staff members treating burn patients
Sampling Method: Non-Probability Sample
Enrollment: 2183 (Estimated)
Dates: Start 2023-01-04 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-15 (Estimated)

PRIMARY OUTCOMES:
Examine the relationships between clinician perceptions of feasibility, acceptability, intention to use, and the actual use of acute burn teleconsultation. | 4 years
  The study team will look at the differences in opinions between the Aim 1 and 2 interviews and surveys as well as the referral numbers being collected and compare that to the Aim 3 data from interviews and surveys as well as actual referral data to see if there is an increase in the use of telemedicine.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - UCI Health Regional Burn Center, Orange, California
  - Massachusetts General Hospital Sumner Redstone Burn Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Regions Hospital Burn Center, Saint Paul, Minnesota

IPD SHARING:
Plan to Share IPD: No